CLINICAL TRIAL: NCT02273167
Title: A Multicenter Randomized Parallel Group Phase III Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of NER1006 (a Low Volume Bowel Cleansing Solution) Versus MOVIPREP Using 2-Day Split-Dosing and 1-Day Morning Split-Dosing Regimen in Adults.
Brief Title: Multicenter Randomized Parallel Group Phase III Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of NER1006 Versus MOVIPREP® Using 2-Day Split-Dosing and 1-Day Morning Split-Dosing Regimen in Adults.
Acronym: MORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NER1006-02/2014 (MORA)
Record Dates: First submitted 2014-10-16; First posted 2014-10-23 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colon Cleansing
MeSH Terms: conditions — Colorectal Neoplasms | interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NER1006, 2-Day Split-Dosing (Experimental): NER1006: 2-Day Split-Dosing Regimen (to commence in the evening of the day before colonoscopy).
  Interventions: Drug: NER1006, 2-Day Split-Dosing
- NER1006,1-Day Morning Split-Dosing (Experimental): NER1006: 1-Day Morning Split-Dosing Regimen (to commence in the morning of the day of colonoscopy).
  Interventions: Drug: NER1006,1-Day Morning Split-Dosing
- MOVIPREP, 2-Day Split-Dosing (Active Comparator): MOVIPREP®: 2-Day Split-Dosing Regimen (to commence in the evening of the day before colonoscopy).
  Interventions: Drug: MOVIPREP, 2-Day Split-Dosing

INTERVENTIONS:
Drug: NER1006, 2-Day Split-Dosing — The subject will self-administer the first dose of the assigned investigational product in the evening prior to the scheduled colonoscopy and take mandatory additional clear fluid. Subject will take the second dose together with mandatory additional clear fluids on the morning of the colonoscopy.
  Arms: NER1006, 2-Day Split-Dosing
Drug: NER1006,1-Day Morning Split-Dosing — The subject will self-administer the first dose of the investigational product on the morning of the colonoscopy and take mandatory additional clear fluid.
  After a 1-2 hour break the subject will self-administer the second dose plus additional clear mandatory fluid.
  Arms: NER1006,1-Day Morning Split-Dosing
Drug: MOVIPREP, 2-Day Split-Dosing — The subject will self-administer the first dose of the assigned investigational product in the evening prior to the scheduled colonoscopy and take recommended additional clear fluid. Subject will take the second dose together with recommended additional clear fluids on the morning of the colonoscopy.
  Arms: MOVIPREP, 2-Day Split-Dosing

SUMMARY:
This study evaluates the efficacy, safety and tolerability of NER1006 versus MOVIPREP in adult patients requiring bowel cleansing prior to any procedure that requires a clean bowel, using a 2-Day evening/morning Split-Dosing and 1-Day morning only Split-Dosing regimens. Approximately 810 patients will be randomised with the aim of achieving a minimum of 245 patients in each of the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent.
* Male and female outpatients and inpatients aged: ≥18 to ≤85 years undergoing a screening, surveillance or diagnostic colonoscopy.
* Females of child-bearing potential must have a negative pregnancy test at Screening and at Visit 2 and must be practising one of the following methods of birth control and agree to continue with the regimen throughout the study period (unless postmenopausal or surgically sterile, or whose sole sexual partner has had a successful vasectomy): Oral, implantable, or injectable contraceptives (for a minimum of three months before study entry) in combination with a condom; Intrauterine device in combination with a condom; Double barrier method (condom* and occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository).
* Willing and able to complete the entire study and to comply with instructions.

Exclusion Criteria:

* Patients with past history within last 12 months or current episode of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Patients with ongoing severe acute Inflammatory Bowel Disease.
* Patients who have had previous significant gastrointestinal surgeries, including colonic resection, sub-total colectomy, abdomino-perineal resection, de-functioning colostomy, Hartmann's procedure and de-functioning ileostomy or other similar surgeries involving structure and function of the small or large colon.
* Regular use of laxatives or colon motility altering drugs in the last month (i.e. more than 2-3 times per week) and/or laxative use within 72 hours prior to administration of the preparation.
* Patients with active intestinal bleeding episodes or with a clinically significant low hemoglobin level <9 g/dL for women and <11 g/dL for men at screening.
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Known phenylketonuria.
* Known hypersensitivity to polyethylene glycols, ascorbic acid and sulfates (not including sulfa-based products) or any other component of the study drug or comparator
* Past history within the last 12 months or evidence of any on-going clinically relevant electrocardiogram (ECG) abnormalities (e.g. arrhythmias).
* History of uncontrolled hypertension with systolic blood pressure >170 mmHg and diastolic blood pressure >100 mmHg.
* Patients with cardiac insufficiency NYHA grades III or IV.
* Patients with severe renal insufficiency (i.e. with GFR, <30 mL/min/1.73m2).
* Patient with serum albumin <3.4 g/dL.
* Patients with liver disease of grades B and C according to the Child Pugh classification.
* Patients suffering from dehydration at screening as evaluated by the Investigator from physical examination and laboratory investigations.
* Patients with clinically significant electrolyte abnormalities, whether pre-existing or noted at screening, such as hypernatremia, hyponatremia, hyperphosphatemia, hypermagnesemia, hypokalemia, hypocalcaemia dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.
* Patients with any other clinically significant hematological parameters including coagulation profile at screening.
* Patients with impaired consciousness that might predispose them to pulmonary aspiration.
* Patients undergoing colonoscopy for foreign body removal and/or decompression.
* Patients who are pregnant or lactating, or intending to become pregnant during the study.
* Clinically relevant findings on physical examination based on the Investigator's judgment.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Concurrent participation in an investigational drug or device study or participation within three months of study entry.
* Patients who are ordered to live in an institution on court or authority order

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raf Bisschops, MD, Principal Investigator — UZ Leuven
Locations (29):
- Belgium (4):
  - AZ Sint-Lucas, Bruges
  - UZ Ghent, Ghent
  - UZ Leuven, Leuven
  - CHC- Clinique Saint-Joseph, Liège
- France (2):
  - Hôpital Avicenne- Service de Gastro-Entérologie, Bobigny
  - Hôpital Hotel-Dieu, Nantes
- Germany (3):
  - Kliniken Essen-Mitte; Abteilung für Gastroenterologie, Essen
  - Klinikum der Friedrich Schiller Universität Jena, Jena
  - Praxis für Innere Medizin, Gastroenterologie und Allg. Medizin, Ludwigshafen
- Italy (5):
  - A.O.U. di Bologna - Policlinico S. Orsola-Malpighi, Bologna
  - Ospedale Valduce U.O. Gastroenterologia e Endoscopia, Como
  - P.O. Maresca OORR Area Vesuviana ASL, Naples
  - Centro di Riferimento Oncologico (C.R.O.) S.O.C Gastroenterologia, Pordenone
  - Pol. Univ. A. Gemelli U.O. di Endoscopia Digestiva Chirurgica, Roma
- Poland (6):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Gabinet Internistyczny dr n. med. Krzysztof Janik, Częstochowa
  - NZOZ Centrum Medyczne-Szpital Swietej Rodziny, Lodz
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych, Warsaw
  - Robert Petryka Gabinet Internistyczny, Warsaw
  - Lexmedica Durbajlo Hanna, Wroclaw
- Spain (5):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Ramon y Cajal - Ctra. De Colmenar km. 9, 100, Madrid
- United Kingdom (4):
  - Lothian Health Board, Edinburgh
  - Borders General Hospital, Melrose
  - Royal Shrewsbury Hospital, Shrewsbury
  - Royal Albert Edward Infirmary Department, Wigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cash BD, Allen C, Poppers DM. Transient alterations in plasma sodium concentrations with NER1006 bowel preparation: an analysis of three phase III, randomized clinical trials. BMC Gastroenterol. 2022 Sep 5;22(1):412. doi: 10.1186/s12876-022-02484-7. PMID 36064325
- [Derived] Bisschops R, Manning J, Clayton LB, Ng Kwet Shing R, Alvarez-Gonzalez M; MORA Study Group. Colon cleansing efficacy and safety with 1 L NER1006 versus 2 L polyethylene glycol + ascorbate: a randomized phase 3 trial. Endoscopy. 2019 Jan;51(1):60-72. doi: 10.1055/a-0638-8125. Epub 2018 Jul 19. PMID 30025414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial recruited out/in-patients at 29 medical centres in Europe, from October 2014 to June 2015.
Period: Overall Study
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Started | 283 | 283 | 283
Completed | 259 | 260 | 262
Not Completed | 24 | 23 | 21
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 10 | 12 | 11
Not completed — Various | 10 | 9 | 8

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis, 245 per arm, was based on assumed overall cleansing success rates of 90% for both MOVIPREP and NER1006, a non-inferiority margin of 10%, and at least 90% power to demonstrate non-inferiority. The overall number of participants analyzed was based on the modified full analysis set (mFAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing | Total
Number analyzed (Participants) | 283 | 283 | 283 | 849
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 228 | 202 | 209 | 639
  >=65 years | 55 | 80 | 74 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.48) | 56.3 (12.03) | 54.9 (13.21) | 55.2 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 163 | 152 | 454
  Male | 144 | 120 | 131 | 395

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Bowel Cleansing (Overall Colon)
Description: The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). A final HCS grading of A, B, C or D was derived. Grades A and B are classified as successful (i.e. all mucosa could be visualized) and C and D are classified as unsuccessful. Comparison of overall success of cleansing with NER1006 2-Day and 1-Day versus MOVIPREP was evaluated using a non-inferiority study design.
Time Frame: Up to 2 days (from day of first dosing to day of colonoscopy)
Population: The overall number of participants analyzed was based on the mFAS. This included all randomized patients, except any patient who (i) was randomized but subsequently failed to meet entry criteria and (ii) in whom it was confirmed (from their patient diary) that the same patient did not receive any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- MOVIPREP, 2-Day Split-Dosing: MOVIPREP: 2-Day Split-Dosing Regimen (to commence in the evening of the day before colonoscopy).
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Number analyzed (Participants) | 272 | 275 | 275
Participants
  Successful | 238 | 253 | 245
  Failure | 34 | 22 | 30
Statistical Analysis 1: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006, 2-Day Split-Dosing; Hypothesis was to demonstrate non-inferiority (NI) of NER1006 2-Day to MOVIPREP (10% margin). Success rate was no. of patients with successful overall bowel cleansing as proportion of no. of patients in each group. Treatment effect was NER1006 2-Day success rate - MOVIPREP success rate. Hochberg procedure used to control Type I error since there were 2 alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — The confidence limits (CL) were adjusted for multiple comparisons (two alternative primary endpoints): To be declared non-inferior, the primary endpoint must show a difference in success rates of no greater than 10% in favour of MOVIPREP using lower 1-sided 97.5% CL. Calculated using exact Clopper-Pearson CLs. To accommodate the comparison of 2 NER1006 regimens a hierarchical testing approach was used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated; p = 0.055, Fisher Exact — The p-value was adjusted for multiple comparisons (two alternative primary endpoints): To be declared superior, primary endpoint must demonstrate non-inferiority with 1-sided p-value <0.025, the threshold for statistical significance; Difference in success rate = 4.50, 97.5% CI 1-sided [lower limit -4.00]
Statistical Analysis 2: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006,1-Day Morning Split-Dosing; The hypothesis was to demonstrate NI of NER1006 1-Day to MOVIPREP (10% margin). Success rate was number of patients with successful overall bowel cleansing as proportion of number of patients in each group. Treatment effect was NER1006 1-Day success rate - MOVIPREP success rate. A Hochberg procedure was used to control Type I error since there were two alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — The CLs were adjusted for multiple comparisons (2 alternative primary endpoints): To be declared non-inferior, the primary endpoint must show a difference in success rates of no greater than 10% in favour of MOVIPREP using lower 1-sided 97.5% CLs. Calculated using exact Clopper-Pearson confidences limits. To accommodate the comparison of two NER1006 regimens a hierarchical testing approach will be used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated; p = 0.328, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in success rate = 1.59, 97.5% CI 1-sided [lower limit -6.91]

2. Primary Outcome: Number of Patients With 'Excellent Plus Good' (Highly Effective) Bowel Cleansing (Colon Ascendens)
Description: The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). Highly effective cleansing in the colon ascendens corresponded to scores 3 (Good) or 4 (Excellent) of the HCS. Adequate plus failure of cleansing corresponded to score 0-2. Comparison of 'Excellent plus good' cleansing of the colon ascendens using NER1006 2-Day and 1-Day versus MOVIPREP was evaluated using a non-inferiority study design.
Time Frame: Up to 2 days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Number analyzed (Participants) | 272 | 275 | 275
Participants
  Excellent plus good | 41 | 87 | 93
  Adequate plus failure | 231 | 188 | 182
Statistical Analysis 1: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006, 2-Day Split-Dosing; Hypothesis was to demonstrate NI of NER1006 2-Day to MOVIPREP (10% margin). Success rate was no. of patients with highly effective cleansing of the colon ascendens as proportion of no. of patients in each group. Treatment effect was NER1006 2-Day success rate - MOVIPREP success rate. Hochberg procedure was used to control Type I error since there were 2 alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — Confidence limits (CL) were adjusted for multiple comparisons (2 alternative primary endpoints): To be declared non-inferior the primary endpoint must show a difference in success rates of no greater than 10% in favour of MOVIPREP using lower 1-sided 97.5% CLs. Calculated using exact Clopper-Pearson CLs. To accommodate the comparison of two NER1006 regimens a hierarchical testing approach will be used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in excellent plus good rate = 16.56, 97.5% CI 1-sided [lower limit 8.11]
Statistical Analysis 2: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006,1-Day Morning Split-Dosing; Hypothesis was to demonstrate NI of NER1006 1-Day to MOVIPREP (10% margin). Success rate was no. of patients with highly effective cleansing of the colon ascendens as proportion of no. of patients in each group. Treatment effect was NER1006 1-Day success rate - MOVIPREP success rate. Hochberg procedure was used to control Type I error since there were 2 alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — The confidence limits (CLs) were adjusted for multiple comparisons (2 alternative primary endpoints): To be declared non-inferior the primary endpoint must show a difference in success rates of no greater than 10% in favour of MOVIPREP using lower 1-sided 97.5% CLs. Calculated using exact Clopper-Pearson CLs. To accommodate the comparison of 2 NER1006 regimens a hierarchical testing approach was used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated; p < 0.001, Fisher Exact — The p-value was adjusted for multiple comparisons (2 alternative primary endpoints): To be declared superior, primary endpoint must demonstrate non-inferiority with 1-sided p-value <0.025, the threshold for statistical significance; Difference in excellent plus good rate = 18.74, 97.5% CI 1-sided [lower limit 10.32]

3. Secondary Outcome: Adenoma Detection Rate (Colon Ascendens)
Description: Comparison of the number of patients with at least one adenoma detected in the colon ascendens when NER1006 2-Day and 1-Day is used for bowel cleansing versus MOVIPREP. Adenoma detection rate (ADR) defined as the number of patients with at least one adenoma in the colon ascendens.
Time Frame: Up to 2 days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Number analyzed (Participants) | 272 | 275 | 275
Participants
  Patients with no adenomas detected | 250 | 243 | 243
  Patients with at least one adenoma detected | 22 | 32 | 32
Statistical Analysis 1: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006, 2-Day Split-Dosing; If at least one of the alternative primary endpoints was met, then key secondary endpoints for the same colon region as met by the primary endpoint were evaluated hierarchically in a pre-specified order. The difference in ADR was calculated as NER1006 2-Day rate - MOVIPREP rate using 1-sided 97.5% confidence limits. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint met non-inferiority. This procedure ensured overall Type I error control at 2.5% 1-sided; Test type: Non-Inferiority or Equivalence — To be declared non-inferior, the key secondary endpoint must show a difference in rates of no greater than 10% in favor of MOVIPREP using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.106, Fisher Exact — To be declared superior, the key secondary endpoint must demonstrate non-inferiority and show a significant advantage for NER1006 2-Day relative to MOVIPREP with 1-sided p-value <0.025, the threshold for statistical significance; Difference in ADR = 3.55, 95% CI 2-sided [-4.80 to 12.00]
Statistical Analysis 2: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006,1-Day Morning Split-Dosing; If at least one of the alternative primary endpoints was met, then key secondary endpoints for the same colon region as met by the primary endpoint were evaluated hierarchically in a pre-specified order. The difference in ADR was calculated as NER1006 1-Day rate - MOVIPREP rate using 1-sided 97.5% confidence limits. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint met non-inferiority. This procedure ensured overall Type I error control at 2.5% 1-sided; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.106, Fisher Exact — To be declared superior, the key secondary endpoint must demonstrate non-inferiority and show a significant advantage for NER1006 1-Day relative to MOVIPREP with 1-sided p-value <0.025, the threshold for statistical significance; Difference in ADR = 3.55, 95% CI 2-sided [-4.80 to 12.00]

4. Secondary Outcome: Adenoma Detection Rate (Overall Colon)
Description: Comparison of the number of patients with at least one adenoma detected in the overall colon when NER1006 2-Day and 1-Day is used for bowel cleansing versus MOVIPREP. Adenoma detection rate (ADR) defined as the number of patients with at least one adenoma in the overall colon.
Time Frame: Up to 2 days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Number analyzed (Participants) | 272 | 275 | 275
Participants
  Patients with no adenomas detected | 199 | 202 | 199
  Patients with at least one adenoma detected | 73 | 73 | 76
Statistical Analysis 1: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006, 2-Day Split-Dosing; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.569, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Difference in ADR = -0.29, 95% CI 2-sided [-8.74 to 8.02]
Statistical Analysis 2: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006,1-Day Morning Split-Dosing; [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.455, Fisher Exact — [p-value comment as in outcome 3, analysis 2]; Difference in ADR = 0.80, 95% CI 2-sided [-7.65 to 9.11]

5. Secondary Outcome: Polyp Detection Rate (Colon Ascendens)
Description: Comparison of the number of patients with at least one polyp detected in the colon ascendens when NER1006 2-Day and 1-Day is used for bowel cleansing versus MOVIPREP. Polyp detection rate (PDR) defined as the number of patients with at least one polyp in the colon ascendens.
Time Frame: Up to 2 days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Number analyzed (Participants) | 272 | 275 | 275
Participants
  Patients with no polyps detected | 228 | 211 | 224
  Patients with at least one polyp detected | 44 | 64 | 51
Statistical Analysis 1: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006, 2-Day Split-Dosing; If at least one of the primary endpoints were met, then key secondary endpoints were evaluated hierarchically in a pre-specified order. Non-inferiority was concluded if the 1-sided 97.5% confidence limit difference in proportion of events between 2 groups excluded a 10% or greater difference was in favor of MOVIPREP. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint had at least met non-inferiority; Test type: Non-Inferiority or Equivalence — To accommodate the comparison of two NER1006 regimens, a hierarchical testing approach was used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated. Difference in Polyp Detection Rate in the colon ascendens was calculated as NER1006 2-Day rate - MOVIPREP rate (10% margin) determined using exact Clopper-Pearson confidence limits; p = 0.024, Fisher Exact; Difference in PDR = 7.10, 95% CI 2-sided [-1.41 to 15.47]
Statistical Analysis 2: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006,1-Day Morning Split-Dosing; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — To accommodate the comparison of two NER1006 regimens, a hierarchical testing approach was used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated. Difference in Polyp Detection Rate in the colon ascendens was calculated as NER1006 rate - MOVIPREP rate (10% margin) determined using exact Clopper-Pearson confidence limits. Non-inferiority of NER1006 1-Day to MOVIPREP was proven; p = 0.268, Fisher Exact — Superiority of NER1006 1-Day to MOVIPREP not demonstrated statistically; Difference in PDR = 2.37, 95% CI 2-sided [-6.12 to 10.82]

6. Secondary Outcome: Polyp Detection Rate (Overall Colon)
Description: Comparison of the number of patients with at least one polyp detected in the overall colon when NER1006 is used for bowel cleansing versus number detected when MOVIPREP is used. PDR defined as the number of patients with at least one polyp in the overall colon.
Time Frame: Up to 2 days (from day of first dosing to day of colonoscopy)
Population: The overall number of participants analysed is based on the mFAS. This included all randomized patients except those patients who (i) were randomized but subsequently failed to meet entry criteria and (ii) in whom it was confirmed (from their patient diary) that the same patient did not receive any study drug (n=822).
Measure: Number; unit: Participants
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Number analyzed (Participants) | 272 | 275 | 275
Participants
  Patients with no polyps detected | 151 | 154 | 151
  Patients with at least one polyp detected | 121 | 121 | 124
Statistical Analysis 1: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006, 2-Day Split-Dosing; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — To accommodate the comparison of two NER1006 regimens, a hierarchical testing approach was used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated. Difference in Polyp Detection Rate in the overall colon was calculated as NER1006 rate - MOVIPREP rate (10% margin) determined using exact Clopper-Pearson confidence intervals; p = 0.579, Fisher Exact; Difference in PDR = -0.49, 95% CI 2-sided [-8.85 to 8.00]
Statistical Analysis 2: Comparison: MOVIPREP, 2-Day Split-Dosing vs NER1006,1-Day Morning Split-Dosing; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — To accommodate the comparison of two NER1006 regimens, a hierarchical testing approach was used whereby NER1006 2-Day was assessed first and, if successful, then NER1006 1-Day was evaluated. Difference in Polyp Detection Rate in the overall colon was calculated as NER1006 1-Day rate - MOVIPREP rate (10% margin) determined using exact Clopper-Pearson confidence limits; p = 0.478, Fisher Exact; Difference in PDR = 0.61, 95% CI 2-sided [-7.78 to 9.09]

ADVERSE EVENTS:
Time Frame: Afternoon of Day 1 (first dose) to Day 9 (final clinic visit)
Description: Treatment Emergent AEs. Safety analyses were based on the safety population, which included all randomized patients whom it could not be ruled out (from their patient diary) that they received study drug at least once (n=794).
Arm/Group | MOVIPREP, 2-Day Split-Dosing | NER1006, 2-Day Split-Dosing | NER1006,1-Day Morning Split-Dosing
Serious Adverse Events (participants affected / at risk) | 0/263 | 2/262 | 0/269
Other Adverse Events (participants affected / at risk) | 31/263 | 41/262 | 49/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOVIPREP, 2-Day Split-Dosing (N=263) | NER1006, 2-Day Split-Dosing (N=262) | NER1006,1-Day Morning Split-Dosing (N=269)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOVIPREP, 2-Day Split-Dosing (N=263) | NER1006, 2-Day Split-Dosing (N=262) | NER1006,1-Day Morning Split-Dosing (N=269)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9) | 15 (16) | 14 (14)
Vomiting (Gastrointestinal disorders) | 3 (3) | 11 (11) | 18 (18)
Fatigue (General disorders) | 5 (5) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 4 (4) | 0 (0) | 1 (1)
Thirst (General disorders) | 2 (2) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Imputation of failure occurred in 4% of patients. This strict analytical approach reduced the cleansing success rates for both treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No